CLINICAL TRIAL: NCT01765673
Title: Passy-Muir Swallowing Self Training Device to Enhance Recovery Post Stroke
Brief Title: The Passy Muir Swallowing Self Training Device
Acronym: PMSST
Status: Completed | Type: Observational
Sponsor: James Madison University (Other)
Collaborators: Passy Muir Inc. (Industry)
Responsible Party: Principal Investigator, Christy Ludlow, Professor, James Madison University
Other Study IDs: R43DC012754 (NIH)
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-09

CONDITIONS: Oropharyngeal Dysphagia
Keywords: Swallowing; Stroke; Sensory stimulation; Home based therapy; Head and Neck Cancer
MeSH Terms: conditions — Deglutition Disorders; Stroke; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vibrotactile Stimulation in Dysphagia: A Vibrotactile stimulation device will be evaluated in patients with chronic moderate to severe dysphagia for more than 6 months post onset due to stroke or following radiation treatment for head and neck cancer to assess which frequency, mode, pressure characteristics are most helpful in increasing the rate of swallowing, increasing the urge to swallow, assisting with the initiation of swallowing and not affecting discomfort.
  Interventions: Device: Vibrotactile stimulation

INTERVENTIONS:
Device: Vibrotactile stimulation — Comparison of the effects of different vibratory characteristics on the frequency of swallowing, time of initiation of swallowing with stimulation and urge to swallow. Will compare frequency of vibration, mode of vibration, pressure of device against neck, and duration of vibration. Each session will last no more than 1 hour with short breaks. Each participant can volunteer for up to three nonconsecutive sessions.
  Other Names: Passy Muir Swallowing Serlf Trainer

SUMMARY:
This is a device evaluation study to determine the optimal stimulation characteristics for using vibrotactile stimulation as a sensory triggering device for self retraining in patients with chronic moderate to severe dysphagia. Stimulation characteristics to be tested are frequency of vibration, pressure between the device and the skin, mode of vibration (pulsed or continuous).

DETAILED DESCRIPTION:
Participants were recruited who had chronic moderate to severe dysphagia following stroke or radiation treatment for head and neck cancer. Their frequency of swallowing was transduced with an accelerometer placed on the skin over the thyroid cartilage and inductive plethysmography bands placed over the rib cage and abdomen. When laryngeal elevation coincided with respiratory apnea a swallow was marked. Five different motor frequencies were evaluated to determine their effect on participants frequency of swallowing (swallows per minute). Frequencies were 30, 70, 110, and 150 Hz and a combination of 70 and 110 Hz. For each vibratory frequency the number of swallows per minute occurring during stimulation was compared with sham when the participant was wearing the device but the motor was not turned on. The frequency fo swallowing during stimulation was compared with the frequency of swallowing between stimulations. Visual analogue ratings of the urge to swallow and discomfort were also measured after each condition. Other parameters were the pressure between the motor and the skin (0, 2, 4, and 6 kPa) and swallow initiation time when stimulation was on and when it was not. Swallowing frequency with continuous versus pulsed stimulation was also compared.

ELIGIBILITY:
Inclusion Criteria:

* Stroke or post radiation for the treatment of head and neck cancer
* Dysphagia with a score of 2 or greater on the Penetration/Aspiration Scale OR a Mann Assessment of Swallowing Ability ordinal risk rating of "probable" or "definite"

Exclusion Criteria:

* Neck injury
* Epilepsy
* Neurological disorder other than stroke
* Psychiatric illness other than depression
* Uncontrolled gastroesophageal reflux disease
* Inability to communicate secondary to significant speech or language problems
* Inability to maintain alertness for 1 hour
* Significant health concerns that would put the participant at risk

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have swallowing problems secondary to a stroke or following radiation for the treatment of head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-01-01; Primary Completion 2016-02-22 (Actual); Study Completion 2016-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christy L Ludlow, PhD, Principal Investigator — James Madison University
Locations (1):
- James Madison University and Rockingham Memorial Hospital, Harrisonburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Theurer JA, Bihari F, Barr AM, Martin RE. Oropharyngeal stimulation with air-pulse trains increases swallowing frequency in healthy adults. Dysphagia. 2005 Fall;20(4):254-60. doi: 10.1007/s00455-005-0021-1. PMID 16633868
- [Result] Theurer JA, Czachorowski KA, Martin LP, Martin RE. Effects of oropharyngeal air-pulse stimulation on swallowing in healthy older adults. Dysphagia. 2009 Sep;24(3):302-13. doi: 10.1007/s00455-009-9207-2. Epub 2009 Apr 24. PMID 19390893

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 13 enrolled, 1 did not pass cognitive testing and did not participate in the study
Period: Overall Study
Arm/Group | Vibrotactile Stimulation in Dysphagia
Started | 12
Completed | 11
Not Completed | 1
Not completed — No transportation for 2nd/3rd visits | 1

BASELINE CHARACTERISTICS:
Population: One of the 13 participants who was consented did not qualify and could not participate. The remaining 12 had severe chronic dysphagia unable to take nourishment by mouth. One of the 12 , 1 was not able to travel for the 2nd or 3rd visit and therefore only partial data are available on the 12 participants.
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Swallow Frequency 30 Hz
Description: Change in number of swallows per minute during stimulation minus swallows per minute during sham (wearing the device but no stimulation)
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in swallows/min
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in swallows/min | 0.512 (1.358)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.218, paired t test

2. Primary Outcome: Change in Swallow Frequency 70 Hz
Description: as for outcome 1
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in Swallows/min
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in Swallows/min | 0.747 (0.924)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.017, paired t test

3. Primary Outcome: Change in Swallow Frequency 110 Hz
Description: as for outcome 1
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in swallows/min
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in swallows/min | 0.849 (1.102)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.022, paired t test

4. Primary Outcome: Change in Swallow Frequency 150 Hz
Description: as for outcome 1
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in swallows/min
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in swallows/min | 0.110 (1.033)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.719, paired t test

5. Primary Outcome: Change in Swallowing Frequency 70 & 110 Hz
Description: as for outcome 1
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in swallows/min
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 11
Change in swallows/min | 0.246 (0.967)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.418, paired t test

6. Secondary Outcome: Change in Urge to Swallow After 30 Hz Stimulation
Description: At the end of each stimulation session participants marked on a visual analogue scale (VAS) their perceived urge to swallow between a minimum of 1 with no urge to swallow and a maximum of 100 which is the highest urge to swallow possible. The Change in perceived urge to swallow when stimulation was presented minus the perceived urge to swallow following no stimulation was computed.
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in VAS Urge to Swallow
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in VAS Urge to Swallow | 18.83 (27.679)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.038, paired t test

7. Secondary Outcome: Change in Urge to Swallow 70 Hz
Description: as for outcome 6
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in VAS Urge to Swallow
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in VAS Urge to Swallow | 13.167 (24.207)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.086, paired t test

8. Secondary Outcome: Change in VAS Urge to Swallow 110 Hz
Description: as for outcome 6
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in VAS Urge to Swallow
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in VAS Urge to Swallow | 12.75 (29.394)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.16, paired t test

9. Secondary Outcome: Change in VAS Urge to Swallow 150 Hz
Description: as for outcome 6
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in VAS Urge to Swallow
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in VAS Urge to Swallow | 14.75 (23.437)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.052, paired t test

10. Secondary Outcome: Change in VAS Urge to Swallow 70 & 110 Hz
Description: as for outcome 6
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in VAS Urge to Swallow
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 11
Change in VAS Urge to Swallow | 2.273 (33.589)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.827, paired t test

11. Secondary Outcome: Change in Discomfort Level 30 Hz
Description: At the end of each stimulation session participants marked on a visual analogue scale (VAS) their perceived discomfort between a minimum of 1 with no discomfort and a maximum of 100 which is the highest discomfort possible. The Change in perceived discomfort when stimulation was presented minus the perceived discomfort following no stimulation was computed.
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in discomfort
Groups:
- Vibrotactile Stimulation in Dysphagia: Vibrotactile stimulation: Comparison of the effects of different vibratory characteristics on the frequency of swallowing, time of initiation of swallowing with stimulation and urge to swallow and discomfort. Will compare frequency of vibration, mode of vibration, pressure of device against neck, and duration of vibration. Each session will last no more than 1 hour with short breaks. Each participant can volunteer for up to three nonconsecutive sessions.
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in discomfort | 2.750 (5.083)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.088, paired t test

12. Secondary Outcome: Change in Discomfort 70 Hz
Description: as for outcome 11
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in discomfort
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in discomfort | 5.25 (11.825)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.152, paired t test

13. Secondary Outcome: Change in Discomfort 110 Hz
Description: as for outcome 11
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in discomfort
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in discomfort | 4.083 (11.12)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.229, paired t test

14. Secondary Outcome: Change in Discomfort 150 Hz
Description: as for outcome 11
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in discomfort
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in discomfort | 5.583 (11.493)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.121, paired t test

15. Secondary Outcome: Change in Discomfort 70 & 110 Hz
Description: as for outcome 11
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in discomfort
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 11
Change in discomfort | 5.273 (13.92)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.239, paired t test

16. Secondary Outcome: Change in Swallowing Frequency 2 kPa
Description: The pressure between the neck band and the skin was set and the changes in swallowing frequency was compared between pressure between increased pressure and no pressure condition
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in Swallow/min
Groups:
- Vibrotactile Stimulation in Dysphagia: Vibrotactile stimulation: Comparison of the effects of different vibratory characteristics on the frequency of swallowing, time of initiation of swallowing with stimulation and urge to swallow and discomfort. Will also compare frequency of vibration, mode of vibration, pressure of device against neck, and duration of swallow initiation. Each session will last no more than 1 hour with short breaks. Each participant can volunteer for up to three nonconsecutive sessions.
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in Swallow/min | 1.417 (1.975)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.03, paired t test

17. Secondary Outcome: Change in Swallow Frequency 4 kPa
Description: as for outcome 16
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in swallows/min
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in swallows/min | 2.0 (3.411)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.067, paired t test

18. Secondary Outcome: Change in Swallow Frequency 6 kPa
Description: The pressure between the neck band and the skin was set and the changes in swallowing frequency was compared between increased pressure and no pressure condition
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: Change in swallows/min
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 12
Change in swallows/min | 1.5 (5.885)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.396, paired t test

19. Secondary Outcome: Percent Change in Swallow Frequency Pulse vs Continuous
Description: Percent Change= [(Number of swallows per minute from continuous stimulation -number of swallows per minute during pulsed stimulation) / number of swallows per minute during pulsed stimulation] X 100
Time Frame: During one session within one hour
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 10
percent change | 37.5 (126.519)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.373, paired t test

20. Secondary Outcome: Change in Swallow Initiation Time
Description: Change in swallow initiation time (ms) from swallow reaction time during vibrotactile stimulation minus reaction time with sham (no) stimulation
Time Frame: During one session within 1 hour
Measure: Mean (Standard Deviation); unit: millisseconds
Groups:
- Vibrotactile Stimulation in Dysphagia: Vibrotactile stimulation: Comparison of the effects of different vibratory characteristics on the frequency of swallowing, time of initiation of swallowing with stimulation and urge to swallow and discomfort. Will compare frequency of vibration, mode of vibration, pressure of device against neck, and swallow initiation time during vibration with no vibration. Each session will last no more than 1 hour with short breaks. Each participant can volunteer for up to three nonconsecutive sessions.
Arm/Group | Vibrotactile Stimulation in Dysphagia
Number analyzed (Participants) | 8
millisseconds | 372 (3092)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation in Dysphagia; Test type: Other; p = 0.744, paired t test

ADVERSE EVENTS:
Time Frame: while enrolled in the study, usually 1 month maximum
Arm/Group | Vibrotactile Stimulation in Dysphagia
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Recruitment was lower than anticipated, we were only able to recruit 12 participants rather than the 15 needed Participants found it burdensome to travel to the testing facility when there was no possible benefit to them for participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2013-10-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT01765673/ICF_000.pdf
  • Study Protocol (2013-10-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT01765673/Prot_001.pdf